CLINICAL TRIAL: NCT03148197
Title: Changes Over Time in the Gut Microbiota of High-risk Hematological Patients Undergoing Allogeneic Stem Cell Transplantation (COLLECT)
Brief Title: Changes in the Gut Microbiota of Patients Undergoing Allogeneic Stem Cell Transplantation (COLLECT)
Acronym: COLLECT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Cologne (Other)
Responsible Party: Principal Investigator, Maria J.G.T. Vehreschild, PD MD, University of Cologne
Other Study IDs: COLLECT
Record Dates: First submitted 2017-05-08; First posted 2017-05-10 (Actual); Last update posted 2017-07-19 (Actual); Status verified 2017-07

CONDITIONS: Acute Myeloid Leukemia; Graft-versus-host-disease; Allogeneic Hematopoietic Stem Cell Transplantation; Stem Cell Transplant Complications
Keywords: Allogeneic hematopoietic stem cell transplantation; Graft-versus-host-disease; Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Graft vs Host Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: None Retained — PBMCs, plasma, urine and stool samples, retention until analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Admitted for allogeneic HSCT: Patients admitted for performance of an allogeneic HSCT after high dosis chemotherapy.
- First diagnosis AML: Patients admitted with a first diagnosis of an acute myeloid leukemia for chemotherapy. Depending on factors like age or molecular risk profile some of these patients will proceed to allogeneic HSCT.

SUMMARY:
COLLECT is a monocentric, prospective, observational study, which aims to assess the association between changes in the intestinal microbiota and the incidence of gastrointestinal graft-versus-host diseases (GvHD). Patients admitted for performance of an allogeneic hematopoietic stem cell transplantation (HSCT) or patients with a first diagnosis of an acute myeloid leukemia (AML) will be enrolled and stool samples will be analyzed using next-generation sequencing. In addition to stool, blood and urine samples will be collected for cytokine and 3-indoxylsulfate analysis.

Exposure to drugs will not be influenced and remains at the discretion of the treating physician.

DETAILED DESCRIPTION:
Documentation of patient is performed by using the web-based survey platform www.ClinicalSurveys.net which was set up by researchers of the University Hospital of Cologne. This survey platform enables an optimal performance in epidemiological, observational, and interventional trials and is characterized by layered access security and frequent data backup. It has been used for numerous registry and cohort studies with approval of competent authorities and ethics boards.

The following data items of patients with a written informed consent are prospectively documented into our database:

* Demographics
* Chemotherapeutic agents
* Other immunosuppressives
* Radiation treatment
* Antibiotic prophylaxis and treatment
* Bowel movement abnormalities
* HSCT Donor and recipient information
* Status of hematological disease
* Days with neutropenia
* Fever and infectious complications

The following samples of patients with a written informed consent are prospectively collected, stored and analyzed:

* Stool samples (16S rRNA analysis)
* Urine (3-IS analysis)
* Ethylenediaminetetraacetic acid (EDTA) blood samples (PBMCs Fluorescence-activated cell sorting (FACS) analysis)
* Citrate blood samples (cytokine analysis)

ELIGIBILITY:
Inclusion Criteria:

* Age of at least 18 years
* Patients admitted for performance of an allogeneic HSCT OR
* Patients with a first diagnosis of an acute myeloid leukemia
* No contraindication for an allogeneic stem cell transplantation
* Subject is not legally incapacitated
* Written informed consent from the study subject has been obtained

Exclusion Criteria:

* Active inflammatory bowel disease
* Ongoing gastroenteritis at the time of inclusion
* Patient has any other condition that, in the opinion of the investigator, would jeopardize the safety or rights of the patient participating in the study, would make it unlikely for the patient to complete the study, or would confound the results of the study
* Persons with any kind of dependency on the investigator or employed by the sponsor or investigator
* Persons held in an institution by legal or official order

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: university hospital cologne
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2017-07-14 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2019-12-31 (Estimated)

PRIMARY OUTCOMES:
Assessment of the association between changes in the intestinal microbiota and the incidence of gastrointestinal GvHD | 365 days
  Analyse changes over time in the intestinal microbiota using 16S ribosomal ribonucleic acid (rRNA) analysis and assess microbiota diversity.

SECONDARY OUTCOMES:
Assessment of the association between changes in the intestinal microbiota and the incidence of non-relapse mortality | 365 days
  Analyse changes over time in the intestinal microbiota using 16S rRNA analysis and assess microbiota diversity.
Investigation of the influence of antibiotics and other risk factors on microbiota changes within this cohort | 365 days
  Analyse changes over time in the intestinal microbiota using 16S rRNA analysis and assess microbiota diversity.
Analysis of the association of 3-indoxylsulfate 3-IS in urine/blood with observed microbiota changes | 365 days
  3-indoxylsulfate (3-IS) concentration levels will be quantified using liquid chromatography in combination with mass spectrometry.
Assessment of the effect of microbiota dysbiosis on cytokine and lymphocyte profiles | 365 days
  Cytokine analysis will be performed on the collected plasma samples (citrate) using multiplex assays and read on a Luminex100™ platform.

CONTACTS AND LOCATIONS:
Overall Officials: Maria Vehreschild, MD, Principal Investigator — University Hospital of Cologne, Department of Internal Medicine / Infectious Diseases, Cologne, Germany
Locations (1):
- University Hospital of Cologne, Cologne, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Taur Y, Jenq RR, Perales MA, Littmann ER, Morjaria S, Ling L, No D, Gobourne A, Viale A, Dahi PB, Ponce DM, Barker JN, Giralt S, van den Brink M, Pamer EG. The effects of intestinal tract bacterial diversity on mortality following allogeneic hematopoietic stem cell transplantation. Blood. 2014 Aug 14;124(7):1174-82. doi: 10.1182/blood-2014-02-554725. Epub 2014 Jun 17. PMID 24939656
- [Background] Jenq RR, Taur Y, Devlin SM, Ponce DM, Goldberg JD, Ahr KF, Littmann ER, Ling L, Gobourne AC, Miller LC, Docampo MD, Peled JU, Arpaia N, Cross JR, Peets TK, Lumish MA, Shono Y, Dudakov JA, Poeck H, Hanash AM, Barker JN, Perales MA, Giralt SA, Pamer EG, van den Brink MR. Intestinal Blautia Is Associated with Reduced Death from Graft-versus-Host Disease. Biol Blood Marrow Transplant. 2015 Aug;21(8):1373-83. doi: 10.1016/j.bbmt.2015.04.016. Epub 2015 May 11. PMID 25977230
- [Background] Weber D, Oefner PJ, Hiergeist A, Koestler J, Gessner A, Weber M, Hahn J, Wolff D, Stammler F, Spang R, Herr W, Dettmer K, Holler E. Low urinary indoxyl sulfate levels early after transplantation reflect a disrupted microbiome and are associated with poor outcome. Blood. 2015 Oct 1;126(14):1723-8. doi: 10.1182/blood-2015-04-638858. Epub 2015 Jul 24. PMID 26209659